CLINICAL TRIAL: NCT00984191
Title: 99mTechnetium-MIBI SPECT-CT for Pre-operative Evaluation of Cervical Lymph Node Metastasis in Papillary Thyroid Carcinoma; A Pilot Study
Brief Title: Pilot 99mTechnetium-MIBI Single Photon Emission Computed Tomography - Computed Tomography (SPECT-CT) in Papillary Carcinoma (CA) Thyroid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Napadon Tangjaturonrasme, Department of Otolaryngology , Faculty of Medicine , Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NapadonChula_01
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Papillary Thyroid Cancer
Keywords: Papillary thyroid cancer; 99mTechnetium MIBI SPECT CT; preoperative; cervical lymphadenopathy; cervical metastasis
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 99mTc positive (Experimental): 99mTechnetium-MIBI SPECT-CT positive compare : Scan - Pathologic report
  Interventions: Radiation: 99mTc-MIBI SPECT-CT
- 99mTc Negative_Neck dissection (Experimental): 99mTc Negative but have neck dissection indication compare : 99mTc - Pathologic report
  Interventions: Radiation: 99mTc-MIBI SPECT-CT
- 99mTc Negative_No neck dissection (Experimental): 99mTc Negative and No other indication for neck dissection compare : 99mTc - 7. 131I (post-treatment) whole body scan
  Interventions: Radiation: 99mTc-MIBI SPECT-CT

INTERVENTIONS:
Radiation: 99mTc-MIBI SPECT-CT — 99mTc-MIBI SPECT-CT for abnormal cervical lymph node

SUMMARY:
The purpose of this trial is to see if the 99mTechnetium-MIBI SPECT-CT can be a tool for preoperative evaluation of cervical node metastasis in papillary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* papillary thyroid cancer

Exclusion Criteria:

* pregnancy
* Bleeding abnormality
* Prior history of head and neck cancer
* can not perform 99mTechnetium-MIBI SPECT-CT
* can not perform 131I remnant Ablation
* Prior any head and neck surgery within 3 months
* Prior deep neck infection within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Tool Statistic (PPV , NPV , Sensitivity , Specificity , Accuracy ) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Napadon Tangjaturonrasme, Otolaryngologist, Principal Investigator — Department of Otolaryngology , Faculty of Medicine , Chulalongkorn University
Locations (1):
- King Chulalongkorn Hospital, Pathumwan, Bangkok, Thailand